CLINICAL TRIAL: NCT01488227
Title: A Prospective Trial on the Effects of Vitamin D Supplementation on 25(OH)D, Body Composition and Injury in Collegiate Swimmers and Divers
Brief Title: A Prospective Trial on the Effects of Vitamin D Supplementation in Collegiate Swimmers and Divers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Kentucky (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: UL1RR033173 (NIH)
Record Dates: First submitted 2011-11-29; First posted 2011-12-08 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: Vitamin D status in athletes; Vitamin D; 25(OH)D; athletes; body composition; inflammatory markers; illness; injury
MeSH Terms: conditions — Wounds and Injuries | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Experimental): Vitamin D
  Interventions: Dietary Supplement: Vitamin D
- Oil pill (Placebo Comparator): Contains vegetable and soybean oil supplied by Nature Made by Pharmavite LLC located in Northridge, CA and is United States Pharmacopeia (USP) certified.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — 4000 IU of Vitamin D daily for 6 months
  Other Names: Vitamin D by Nature Made by Pharmavite LLC
  Arms: Vitamin D
Dietary Supplement: Placebo — Acts as a control for the Vitamin D intervention
  Other Names: Placebo by Nature Made by Pharmavite LLC
  Arms: Oil pill

SUMMARY:
Objective 1: Determine if Vitamin D supplementation can improve body composition, reduce injuries and illnesses, and improve performance in collegiate swimmers and divers.

Objective 2: Examine how baseline Vitamin D levels predict outcome variables over the course of the intervention period.

DETAILED DESCRIPTION:
The investigators plan to recruit from approximately 45 male and female University of Kentucky Swimmers and Divers, at least 18 years of age in August 2011. Approximately equal numbers of men and women will be recruited. The entire athletic team(s) will be recruited. With a conservative dropout rate of 30%, the investigators final sample size should be approximately 22 participants (per group).Following baseline measures, participants will be randomized to one of two groups (Vitamin D 4000 IU or Placebo control) and monitored over the course of their athletic season. Measurements will be repeated at Midpoint (3 months) and Endpoint (6 months).

Participants will have no recent history of Vitamin D supplementation beyond what is normally found in a multivitamin (400 IUs).

Following the informed consent process a medical history and Vitamin D questionnaire (screenings), and urine pregnancy test (for female athletes) will be administered prior to more invasive baseline testing procedures (blood draw and DXA). A blood draw will then be conducted at baseline, midpoint and endpoint. Collected blood for the purposes of this study will assess Vitamin D status (25(OH)D), parathyroid hormone, ionized calcium, bone turnover markers, and inflammatory cytokines. A Vitamin D lifestyle questionnaire will be administered at all 3 time points and incidence of illness and injury will be documented over 6 months following randomization. DXA measures will only occur at Baseline and Endpoint.

ELIGIBILITY:
Inclusion Criteria:

* University of Kentucky Swimmers and Divers, at least 18 years old.
* No recent history of Vitamin D supplementation beyond 400IU

Exclusion Criteria:

* hormone replacement therapy,
* high dose Vitamin D supplementation,
* history of renal disease or kidney stones,
* organ transplantation,
* sarcoidosis,
* parathyroid disease,
* history of high blood calcium levels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
25(OH)D) | 3 measurement periods over 6 months
  Baseline, Midpoint, and Endpoint measures include a blood draw for 25(OH)D status.

SECONDARY OUTCOMES:
Inflammatory Cytokines | Baseline and Enpoint
  Baselineand Endpoint measures include a blood draw inflammatory cytokines (TNF alpha, IL1-B, IL6)
Bone Turnover Markers | Baseline, Midpoint, Endpoint
  Baseline, Midpoint, and Endpoint measures include a blood draw for bone turnover markers (BSAP, NTx).
DXA Body Composition | Baseline and Endpoint
  Baseline and Endpoint measures include Body Composition measures (DXA) for fat, muscle and bone composition
Vitamin D Lifestyle Survey | Baseline, Midpoint, Endpoint
  Baseline, Midpoint, and Endpoint measures include a behavioral survey for estimating 25(OH)D status (solar exposure, food and other supplemental intake)
injury and illness incidence | 6 months
  We will track injury and illness type and incidence over the course of the 6 month intervention

CONTACTS AND LOCATIONS:
Overall Officials: Maja Redzic, B.S., Study Director — University of Kentucky; Regina M Lewis, B.S., Study Director — University of Kentucky; David T Thomas, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States